CLINICAL TRIAL: NCT04186078
Title: Clinical Characteristics of Patients With Sleep Apnea in Korea: a Prospective Cohort Study
Brief Title: Clinical Characteristics of Patients With Sleep Apnea in Korea
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jaeyoung Cho, Assistant Professor, Seoul National University Hospital
Other Study IDs: 19071511050
Record Dates: First submitted 2019-11-27; First posted 2019-12-04 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For only participants with the informed consent of donating blood, their blood samples (serum, plasma, and buffy coat) will be collected and stored in the Seoul National University Hospital-Human Biobank (SNUH-HUB).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- obstructive sleep apnea (OSA): 5 or more predominantly obstructive respiratory events [obstructive and mixed apneas, hypopneas or respiratory effort-related arousals (RERAs)] per hour of sleep during a PSG or per hour of monitoring (respiratory polygraphy)
- central sleep apnea (CSA): PSG shows all of the following:
  1. 5 or more central apneas and/or central hypopneas per hour of sleep.
  2. The number of central and/or central hypopneas is > 50% of the total number of apneas and hypopneas.
- control: apnea-hypopnea index < 5 per hour of sleep during a PSG or per hour of monitoring (respiratory polygraphy)

SUMMARY:
Sleep-disordered breathing including obstructive sleep apnea (OSA) is an extremely common medical disorder associated with important morbidity. The purpose of this study is to understand the clinical features and course of patients with sleep apnea in Korea. Participants who are suspected of sleep apnea due to symptoms such as snoring, witnessed apneas, waking up with a choking sensation, excessive sleepiness, non-restorative sleep, difficulty initiating or maintaining sleep, fatigue or tiredness, and morning headache will be prospectively recruited at the outpatient clinic of Seoul National University Hospital. After polysomnography (PSG) or respiratory polygraphy, patients with sleep apnea including OSA and central sleep apnea (CSA) will be followed regularly. Participants not having sleep apnea (apnea-hypopnea index < 5/hour) will only have a baseline visit. For only participants with the informed consent of donating blood, their blood samples will be collected and stored in the Seoul National University Hospital-Human Biobank (SNUH-HUB).

ELIGIBILITY:
Inclusion Criteria:

* Participants who are suspected of sleep apnea due to symptoms such as snoring, witnessed apneas, waking up with a choking sensation, excessive sleepiness, non-restorative sleep, difficulty initiating or maintaining sleep, fatigue or tiredness, and morning headache

Exclusion Criteria:

* None

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants who are suspected of sleep apnea due to symptoms such as snoring, witnessed apneas, waking up with a choking sensation, excessive sleepiness, non-restorative sleep, difficulty initiating or maintaining sleep, fatigue or tiredness, and morning headache will be prospectively recruited at the outpatient clinic of Seoul National University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2045-12 (Estimated); Study Completion 2046-12 (Estimated)

PRIMARY OUTCOMES:
The number of participants with adherence to positive airway pressure (PAP) therapy | Median follow up of 2 years
  PAP adherence is defined as the use of PAP therapy for ≥4 h/night on ≥70% of nights

SECONDARY OUTCOMES:
The number of deaths | Median follow up of 15 years
  The number of deaths
The cause of death | Median follow up of 15 years
  The cause of death

OTHER OUTCOMES:
Change of FEV1 and FVC in patients with OSA | Median follow up of 5 years
  Change of forced expiratory volume in 1 s (FEV1) and forced vital capacity (FVC) in patients with OSA

CONTACTS AND LOCATIONS:
Overall Officials: Jaeyoung Cho, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea